CLINICAL TRIAL: NCT02239614
Title: A Phase 1, Randomized, Open-label, Single-center, Study of TDENV-PIV and LAV Dengue Vaccine Platforms as Part of a Heterologous Prime-boost Strategy in Healthy Adults in a Nonendemic Region
Brief Title: TDENV PIV and LAV Dengue Prime-boost Strategy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-13-10; ADVP-003 (Other: Sponsor); WRAIR #2136 (Other: WRAIR)
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Dengue
Keywords: dengue fever; dengue
MeSH Terms: conditions — Dengue | interventions — Aluminum Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: LAV (T=0), PIV (T=28) (Experimental): Tetravalent live-attenuated dengue virus vaccine formulation 17 (TDENV-LAV) reconstituted with 0.7 mL of water-for-injection; administered subcutaneously on day 0 of the study.
  Tetravalent dengue purified inactivated vaccine 4 μg/serotype with alum adjuvant (TDENV-PIV 4 µg + alum adjuvant) administered intramuscularly on day 28 of the study.
  Interventions: Biological: TDENV-LAV; Biological: TDENV-PIV 4 µg + alum adjuvant
- Group 2: PIV (T=0), LAV (T=28) (Experimental): Tetravalent dengue purified inactivated vaccine 4 μg/serotype with alum adjuvant (TDENV-PIV 4 µg + alum adjuvant) administered intramuscularly on day 0 of the study.
  Tetravalent live-attenuated dengue virus vaccine formulation 17 (TDENV-LAV) reconstituted with 0.7 mL of water-for-injection; administered subcutaneously on day 28 of the study.
  Interventions: Biological: TDENV-LAV; Biological: TDENV-PIV 4 µg + alum adjuvant
- Group 3: LAV (T=0), PIV (T=180) (Experimental): Tetravalent live-attenuated dengue virus vaccine formulation 17 (TDENV-LAV) reconstituted with 0.7 mL of water-for-injection; administered subcutaneously on day 0 of the study.
  Tetravalent dengue purified inactivated vaccine 4 μg/serotype with alum adjuvant (TDENV-PIV 4 µg + alum adjuvant) administered intramuscularly on day 180 of the study.
  Interventions: Biological: TDENV-LAV; Biological: TDENV-PIV 4 µg + alum adjuvant
- Group 4: PIV (T=0), LAV (T=180) (Experimental): Tetravalent dengue purified inactivated vaccine 4 μg/serotype with alum adjuvant (TDENV-PIV 4 µg + alum adjuvant) administered intramuscularly on day 0 of the study.
  Tetravalent live-attenuated dengue virus vaccine formulation 17 (TDENV-LAV) reconstituted with 0.7 mL of water-for-injection; administered subcutaneously on day 180 of the study.
  Interventions: Biological: TDENV-LAV; Biological: TDENV-PIV 4 µg + alum adjuvant

INTERVENTIONS:
Biological: TDENV-LAV — 0.5 mL of the post-transfection LAV F17 vaccine
  Other Names: TDENV-LAV F17; Tetravalent dengue live attenuated virus formulation 17
Biological: TDENV-PIV 4 µg + alum adjuvant — 0.5 mL of DENV serotypes 1-4 (4 µg / serotype) in alum adjuvant
  Other Names: Tetravalent dengue virus purified inactivated vaccine with alum adjuvant

SUMMARY:
The potential synergistic effect of administering 2 dengue vaccine candidates that were previously shown to be safe and immunogenic in humans will be evaluated in this study. A prime-boost study of tetravalent dengue virus purified inactivated vaccine (TDENV-PIV) with alum and tetravalent dengue live attenuated virus (TDENV-LAV) vaccine Formulation 17 (F17) will gather data to help better understand the human immune response to dengue vaccination and infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 49 years of age (inclusive) at the time of consent
2. Able to provide written informed consent
3. Healthy as established by medical history and clinical examination before entering into the study
4. Able and willing to comply with the requirements of the protocol (eg, document events in memory aid, return for follow-up visits, etc.)
5. Female subject of non-childbearing potential (non-childbearing potential is defined as having either a current tubal ligation at least 3 months prior to enrollment or a history of a hysterectomy, ovariectomy, or is post-menopause)
6. Female subject is not breastfeeding and agrees not to breastfeed for 3 months after last vaccination
7. Female subject of childbearing potential may be enrolled in the study, if the subject has:

   1. Practiced adequate contraception for 30 days prior to vaccinations, and
   2. A negative urine pregnancy test on each day of vaccination, and
   3. Agreed to continue adequate contraception until 3 months after completion of the vaccination series.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines during the period starting 30 days preceding the first dose of study vaccine and/or planned use during the study period
2. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to the first vaccine dose

   1. For corticosteroids, this will mean prednisone ≥ 20 mg/d or equivalent
   2. Inhaled and topical steroids are allowed
3. Planned administration or administration of a vaccine/product not foreseen by the study protocol during the period starting 14 days before or after each scheduled dose of an investigational product
4. Planned administration of any flavivirus vaccine for the entire study duration
5. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device)
6. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required)
7. Family history of congenital or hereditary immunodeficiency
8. History of, or current, auto-immune disease
9. History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or related to a study procedure
10. Major congenital defects or serious chronic illness
11. History of any neurological disorders or seizures. (except for a childhood febrile seizures)
12. Acute disease and/or fever (oral body temperature ≥ 100.4°F/38.0°C) at the time of enrollment (a subject with a minor illness, ie, mild diarrhea, mild upper respiratory infection, etc, without fever, may be enrolled at the discretion of the investigator)
13. Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests
14. Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the first dose of study vaccine or planned administration during the study period
15. History of chronic alcohol and/or drug abuse
16. Pregnant or breastfeeding female or female planning to become pregnant or planning to discontinue contraceptive precautions
17. A planned move to a location that will prohibit participating in the trial prior to the study end for the participant
18. Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
19. Safety laboratory test results that are outside the acceptable values at screening:

    1. > 110% upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, creatinine, serum urea nitrogen (SUN) and bilirubin (total and direct)
    2. < 100% lower limit of normal (LLN) or > 120% ULN for hemoglobin, hematocrit and platelet count
    3. < 75% LLN or >110% ULN for total white blood cell count (WBC)
20. Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Number of solicited adverse events | 21 days after each vaccination
Number of unsolicited adverse events | 28 days after each vaccination
Number of hematological and biochemistry abnormalities | 7 and 28 days and each vaccination
Number of serious adverse events | Day 208 or day 360
Number of potential immune-mediated diseases | Day 208 or day 360
Number of medically attended adverse events | Day 208 or day 360

SECONDARY OUTCOMES:
Microneutralizing (MN) dengue antibody titers | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MAJ Leyi Lin, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Clinical Trials Center, Walter Reed Army Institute of Research (CTC, WRAIR), Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Lin L, Koren MA, Paolino KM, Eckels KH, De La Barrera R, Friberg H, Currier JR, Gromowski GD, Aronson NE, Keiser PB, Sklar MJ, Sondergaard EL, Jasper LE, Endy TP, Jarman RG, Thomas SJ. Immunogenicity of a Live-Attenuated Dengue Vaccine Using a Heterologous Prime-Boost Strategy in a Phase 1 Randomized Clinical Trial. J Infect Dis. 2021 May 28;223(10):1707-1716. doi: 10.1093/infdis/jiaa603. PMID 32966573